CLINICAL TRIAL: NCT04946435
Title: Evaluating the Effect of Prophylactic Topical Antibiotic Irrigation on Nasal Packing Colonization Following Endoscopic Skull Base Surgery
Brief Title: Topical Antibiotic Prophylaxis for Nasal Packing Post-ESBS
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: We are no longer going to undertake the study.
Sponsor: Carl Snyderman (Other)
Responsible Party: Sponsor-Investigator, Carl Snyderman, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY21040170
Record Dates: First submitted 2021-06-16; First posted 2021-06-30 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Intracranial Pathology

STUDY DESIGN:
Intervention Model Description: Participants will consist of 60 patients undergoing primary or revision endoscopic skull base surgery. The first 30 patients will be assigned to the control group to collect data on common nasal packing colonization and appropriate antibiotic selection for the experimental group. The following 30 patients will be assigned to the experimental group. Immediately following surgery, the control group will receive nasal packing alone and the experimental group will receive nasal packing with antibiotic irrigation.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Drug: Antibiotic Irrigation, and Procedure/Surgery: Nasal Packing (Experimental): Experimental group will receive nasal packing with antibiotic irrigation.
  Interventions: Combination Product: Antibiotic Irrigation
- Procedure/Surgery: Nasal Packing (Active Comparator): Patients will be assigned to the control group to collect data on common nasal packing colonization and appropriate antibiotic selection for the experimental group.
  Interventions: Combination Product: Antibiotic Irrigation

INTERVENTIONS:
Combination Product: Antibiotic Irrigation — The first 30 patients will be assigned to the control group to collect data on common nasal packing colonization and appropriate antibiotic selection for the experimental group. The following 30 patients will be assigned to the experimental group. Immediately following surgery, the control group will receive nasal packing alone and the experimental group will receive nasal packing with antibiotic irrigation

SUMMARY:
This is an interventional study that will examine the effect of prophylactic topical antibiotics on nasal packing colonization following endoscopic skull base surgery.

DETAILED DESCRIPTION:
Following endoscopic skull base surgery (ESBS), nasal packing is used to control bleeding and to support reconstruction but can be a source for possibly infectious colonization. Antibiotic use and selection in ESBS varies largely and topical antibiotics are not routinely employed despite favorable qualities (i.e. direct delivery of high antibiotic concentrations with low adverse systemic effects). The effect of prophylactic topical antibiotics on nasal packing colonization is currently understudied. A larger study is needed to test the validity of the conclusion. Employing a larger sample size undergoing ESBS (which does not directly act on the nasal cavity), the investigators hope to amend the lack of literature evaluating the effect of prophylactic topical antibiotics on nasal packing post-ESBS. THe investigators hope to contribute to the determination of an ideal antibiotic regimen following ESBS, which may be especially beneficial for immunocompromised patients or patients at risk of post-surgery infections such as meningitis. Furthermore, the effect of ESBS on the nasal flora is largely understudied, with limited literature only reporting on the nasal flora following endoscopic sinus surgery (ESS). The investigators hope to also amend the lack of literature exploring the effects of ESBS on the nasal flora, especially long-term effects that may be examined in patients undergoing revision surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary or revision endoscopic skull base surgery
* Sellar or Intracranial pathology

Exclusion Criteria:

* Patients with sinonasal malignancy
* Prior radiation therapy
* Concurrent sinusitis and/or nasal polyposis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Can prophylactic topical antibiotics alter the colonization of nasal packing following endoscopic skull base surgery | 1 year
  The effect of prophylactic topical antibiotics on nasal packing colonization post-endoscopic skull base surgery will be measured using culture analysis. Colonization will be described as type(s) of bacteria.
Can prophylactic topical antibiotics alter the bacterial load of nasal packing following endoscopic skull base surgery | 1 year
  The effect of prophylactic topical antibiotics on the bacterial load of nasal packings post-endoscopic skull base surgery will be measured using culture analysis. Bacterial load will be measured in colony forming units (CFUs).
Which bacteria colonize nasal packing following endoscopic skull base surgery | 1 year
  The bacteria making up the colonization of nasal packing post-endoscopic skull base surgery will be identified using culture analysis.

SECONDARY OUTCOMES:
Does endoscopic skull base surgery later the nasal flora | 1 year
  A secondary endpoint is to determine if ESBS alters the nasal flora. The change in nasal flora after endoscopic skull base surgery will be measured using culture analysis of pre- and post-surgery nasal swabs

OTHER OUTCOMES:
Does nasal packing colonization correlate with causative organisms | 1 year
  The similarities or differences in bacteria colonizing nasal packings post-surgery in the study sample and causing meningitis in previous skull base patients will be investigated using culture analysis and chart review.

CONTACTS AND LOCATIONS:
Overall Officials: Carl Snyderman, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No